CLINICAL TRIAL: NCT07296991
Title: VR Stimulation of Exercise Response in Sedentary Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Alyson Sujkowski, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-23-06-5927; 5R01AG059683-07 (NIH)
Record Dates: First submitted 2025-12-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prolonged Inactivity; Metabolic Syndrome
Keywords: Exercise; metabolic syndrome; insulin resistance; virtual reality
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EX-20 minutes sub max cycling exercise (Active Comparator): 20 minutes cycling exercise
  Interventions: Behavioral: 20 minutes cycling exercise
- VR-virtual reality exercise (Experimental): 20 minutes virtual cycling
  Interventions: Behavioral: Virtual Reality
- VR+: 20 minutes sub max cycling exercise + virtual reality (Active Comparator): 20 minutes cycling exercise + 20 minutes virtual cycling
  Interventions: Behavioral: 20 minutes cycling exercise; Behavioral: Virtual Reality

INTERVENTIONS:
Behavioral: 20 minutes cycling exercise — 20 minutes cycling exercise
  Arms: EX-20 minutes sub max cycling exercise; VR+: 20 minutes sub max cycling exercise + virtual reality
Behavioral: Virtual Reality — 20 minutes virtual cycling
  Arms: VR+: 20 minutes sub max cycling exercise + virtual reality; VR-virtual reality exercise

SUMMARY:
Prolonged sedentary conditions contribute to declining health across human populations and cause significant secondary health consequences for many patients whose illnesses or injuries prevent them from exercising. The investigators have demonstrated that in a small animal fruit fly model, genetic stimulation of neurons that promote adrenergic signaling is sufficient to mimic the benefits of exercise training even in sedentary animals. The investigator's pilot work in humans has confirmed that humans respond to Virtual Reality (VR) stimuli that mimic exercise by increasing heart rate and altering heart rate variability in a way consistent with increased adrenergic activity.

In this study, the investigators will directly test for the first time whether repeated, controlled exposure to VR stimuli that induce adrenergic activity in sedentary humans can produce adaptive changes to protein expression and endurance performance like those produced by actual exercise in pre-diabetic participants with/without hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Equal numbers male and female (32 each)
2. Blood glucose HbA1C: 5.7-6.4% or 100-125 mg/dL
3. BP: systolic<120 and diastolic<80 mmHg, systolic 120-129 mmHg and diastolic <80 mmHg, or systolic >130 mmHg and diastolic >80 mmHg

Exclusion Criteria:

1. BMI>35kg/m2
2. Currently involved in an exercise program or similar activity
3. Taking medications that could affect results, including beta-blockers or SSRIs
4. Demonstrate any form of discomfort with the VR experience through self-reported feelings of anxiety or nausea
5. Alcohol consumption above a minimal level(<2 oz/night)
6. BP: Systolic >160 mmHg and Diastolic >110 mmHg

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose, HbA1C | 10 weeks
  Pre-diabetic patients (Blood glucose 100-125 mg/dL, AbA1C 5.7-6.4%) may see improvement in values post-intervention

SECONDARY OUTCOMES:
10 minute walk time | 10 weeks
  distance walked in 10 minutes is recorded pre- and post- intervention and may improve

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Wessells, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Data from human studies will be shared in aggregate and/or deidentified form at the time of publication and backed up on shared drives among the study personnel according to the terms of the Institutional Review Board and the approved consent forms. Identifying data will be kept in a locked cabinet under supervision of the PI and destroyed at the conclusion of the study